CLINICAL TRIAL: NCT00430573
Title: Placebo-Controlled Evaluation of the Efficacy of D-Cycloserine for Enhancing the Effects of CBT for Substance Use
Brief Title: Efficacy of D-Cycloserine for Enhancing the Effects of CBT for Substance Use
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The investigators failed to recruit participants as originally projected.
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael Otto, Ph.D., Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01 DA017904-S1; R01DA017904 (NIH)
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Substance-Related Disorders
Keywords: cognitive-behavior therapy; d-cycloserine; cognitive enhancer; drug dependence; opiate dependence; exposure; isolated doses of d-cycloserine; isolated doses of matching pill placebo; DCS
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DCS-augmented CBT-IC (Experimental): D-cycloserine-augmented CBT-IC
  Interventions: Drug: D-cycloserine
- Placebo-augmented CBT-IC (Placebo Comparator): Placebo-augmented CBT-IC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — Single dosage of D-cycloserine is given prior to each of 6 sessions of CBT-IC treatment (sessions 5-10)
  Other Names: DCS
  Arms: DCS-augmented CBT-IC
Drug: Placebo — Single dosage of placebo is given prior to each of 6 sessions of CBT-IC treatment (sessions 5-10)
  Arms: Placebo-augmented CBT-IC

SUMMARY:
This study examines whether isolated doses of d-cycloserine enhance the efficacy of an exposure-based cognitive-behavioral treatment for chronic and treatment refractory substance dependence.

DETAILED DESCRIPTION:
This is a placebo-controlled trial of the efficacy of 50mg d-cycloserine or matching pill placebo for enhancing the efficacy of CBT.

ELIGIBILITY:
Inclusion criteria:

The primary selection criteria include women and men between the ages of 18 and 65 who:

1. Meet DSM-IV criteria for opiate dependence,
2. Maintain a stable dose of methadone for two weeks prior to recruitment and:

   * fail to achieve "take-home" status for methadone dosing during at least the first four months of methadone treatment,
   * test positive on at least two toxicology screens for illicit drugs during the month prior to recruitment
   * have never achieved two consecutive toxicology screens free of illicit substances since entering the current treatment episode.
3. Meet study criteria for chronic stress:

   * unemployment criteria, and
   * affective disorder criteria.

Exclusion Criteria:

1. Patients with significantly unstable or uncontrolled medical illness which may interfere with participation in treatment (e.g., patients likely to require hospitalization during the study period).
2. Patients with a psychotic or organic mental disorder according to DSM-IV criteria.
3. Patients receiving medication affecting methadone metabolism (e.g. rifampin).
4. Patients with uncontrolled bipolar disorder as evidenced by meeting current criteria for mania or hypomania or meeting criteria for rapid cycling in the last year (as indicated by structured questioning of all patients meeting criteria for bipolar disorder).
5. Patients unable to complete the informed consent or unable to understand study procedures in the informed consent process.
6. Pregnancy or current alcohol use.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Otto, Ph.D., Principal Investigator — Boston University
Locations (1):
- Habit OPCO, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This pilot study was terminated due to inadequate recruitment. The primary reason was unwillingness to take a study drug (a parent study that did not require randomized drug was likely a factor in this decision).
Pre-assignment Details: 15 people consented to this study but 4 did not meet entry criteria and 1 was loss to follow-up before completing baseline evaluations. 10 participants were randomized and 5 dropped out before taking study drug.
Groups:
- All Randomized Participants: The blind was never broken for the study drug, therefore, results can only be presented aggregated for all randomized participants.
Period: Overall Study
Arm/Group | All Randomized Participants
Started | 10
Completed | 5 (Only 5 took study drug on at least one occasion and 8 completed the baseline ASI.)
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: 10 participants were randomized out of the initial15 who consented to the study
Groups:
- Overall Study Characteristics: All participants who consented to be in the study
Arm/Group | Overall Study Characteristics
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Positive Toxicology Swabs for Illicit Substances
Description: The primary outcome assessment for this study was the percentage of oral toxicology swabs that were positive of illicit substances. Participants completed these swabs at each assessment point, as well as at each study therapy session. Toxicology swabs were supervised by study staff and used oral specimen collection to screen for opiates, methadone, cocaine, benzodiazepines, amphetamines, THC, and barbiturates.
Time Frame: Weekly assessments with summation over three time periods: baseline, treatment (week 12), and follow-up (week 18)
Population: Toxicology swabs were obtained on all 10 randomized participants irrespective of taking study drug. At baseline all 10 had toxicology swabs, at treatment (week 12) 7 had toxicology swabs and at follow-up (week 18) 7 had toxicology swabs.
Measure: Mean (Standard Deviation); unit: percentage of positive toxicology swabs
Groups:
- All Randomized Participants: 10 participants were randomized and 5 dropped out before taking study drug. The blind was never broken for the study drug, Therefore, results can only be presented aggregated for all randomized participants.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 10
percentage of positive toxicology swabs
  Baseline Period | 80.0 (35.0)
  Treatment Period (week12): number analyzed (Participants) | 7
  Treatment Period (week12) | 65.7 (45.8)
  Follow-up Period (week 18): number analyzed (Participants) | 7
  Follow-up Period (week 18) | 59.6 (44.1)

2. Secondary Outcome: Addiction Severity Index (ASI) Drug Use Composite Score
Description: For the drug use composite scores, each of 13 questions about drug use is divided by its maximum answer value and by the total number of questions in the composite. These individual items are then summed, so that possible total scores range from 0 to 1, with higher scores reflecting greater drug use problem severity.
Time Frame: Baseline, Mid Treatment (week 6), End of Treatment (week 12), Follow-up 1 (week 15), Follow-up 2 (week 18)
Population: All randomized participants were asked to complete the ASI irrespective of taking study drug. At least one ASI was completed by 8 of the 10 randomized participants. At baseline 8 completed the ASI and the number of participants at each subsequent time point varied.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Randomized Participants That Completed Baseline ASI: 8 of the 10 randomized participants completed the baseline ASI evaluation.
Arm/Group | Randomized Participants That Completed Baseline ASI
Number analyzed (Participants) | 8
units on a scale
  Baseline | 0.27 (0.14)
  Mid-Treatment (week 6) | 0.19 (0.12)
  Endpoint of Treatment (week 12): number analyzed (Participants) | 6
  Endpoint of Treatment (week 12) | 0.21 (0.13)
  Follow-Up 1 (week 15): number analyzed (Participants) | 4
  Follow-Up 1 (week 15) | 0.30 (0.06)
  Follow-Up 2 (week 18): number analyzed (Participants) | 5
  Follow-Up 2 (week 18) | 0.18 (0.18)

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | All Randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Study was terminated due to low enrollment/adherence with the study drug. 10 participants were randomized, 5 dropped out before taking study drug. The blind was never broken so results can only be presented aggregated for all randomized participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes